CLINICAL TRIAL: NCT01757080
Title: Cardiorespiratory Performance in Diabetic Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Daniella Cunha Brandao, PhD, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: etiene
Record Dates: First submitted 2012-12-04; First posted 2012-12-28 (Estimated); Last update posted 2012-12-28 (Estimated); Status verified 2012-10

CONDITIONS: Diabetics Patients; Hypertensive Patients

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diabetic-hypertensive elderly (Experimental): Biochemical analysis and Cardiorespiratory performance assessment with ergospirometry test
  Interventions: Other: Cardiorespiratory performance assessment with ergospirometry test; Other: Biochemical analysis
- Hypertensive elderly (Active Comparator): Biochemical analysis and Cardiorespiratory performance assessment with ergospirometry test
  Interventions: Other: Cardiorespiratory performance assessment with ergospirometry test; Other: Biochemical analysis

INTERVENTIONS:
Other: Cardiorespiratory performance assessment with ergospirometry test
Other: Biochemical analysis

SUMMARY:
OBJECTIVE: To analyze the influence of lipid control during a cardiorespiratory exercise test in two subgroups. DESIGN: Parallel trial study. PARTICIPANTS: The sample consisted of 40 elderly people, male and female, divided into two groups: 20 hypertensive (G1; 68.50 ±5.85 years) and 20 diabetic-hypertensive (G2; 68.95 ±6.79 years). MEASUREMENTS: Nutritional status; glucose and lipid controls - postprandial glucose (PPG), triglycerides (TG), total cholesterol (TC), low density lipoprotein (LDL-C), very low density lipoprotein (VLDL-C), high density lipoprotein (HDL-C); blood pressure, and cardiorespiratory performance. The significance level was set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* 60-years-old or above
* diagnosis of hypertension and/or T2DM for at least 2 years
* member active of the hypertension and diabetes mellitus program
* be on optimized drug therapy for more than 3 months
* BMI above 22 kg/m²;
* no heart disease
* non-insulin-dependent,
* sedentary according to the International Physical Activity Questionnaire (IPAQ) and
* functionally independent.

Exclusion Criteria:

* ergospirometry interrupted by adaptive,
* hemodynamic, and electrocardiographic complications;
* respiratory exchange ratio (R) lower than 1.0 at the end of exertion,
* VE/VCO2 value higher than 34 in the first anaerobic threshold;
* chronic atrial fibrillation;
* neuromuscular,
* orthopedic,
* peripheral vascular,
* pulmonary diseases;
* myocardial infarction within 6 months;
* orthopedic limitation or musculoskeletal pain.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory exercise test | six months
  To analyze the influence of lipid control during a cardiorespiratory exercise test in two subgroups.

SECONDARY OUTCOMES:
Physical activity level assessment performed with the International Physical Activity Questionnaire (IPAQ) | Six months
  This questionnaire was validated in a Brazilian population and in an interview approach. It contains questions regarding frequency and duration of physical activities, classifying the elderly in four categories: very active, active, irregularly active, and sedentary. The physical activity level was investigated considering two variables: Sedentariness and "Time of moderate intensity activities" (TMIA). The presence of sedentariness was established in those subjects who were classified as sedentary and all other classifications were grouped as absence of sedentariness. The TMIA referred to the time self-reported by the subjects, weekly, in minutes spent in performing moderate intensity activities , calculated according to the answers to questions 2a and 2b from IPAQ, as follows: TMIA = (n days) x (time in min).
Assessment of functional capacity was quantitatively analyzed based on the scores obtained in the Instrumental Activities of Daily Living (IADL). | Six months
  This scale has as maximum score 27 points, with the following classification: (27-26 points), partially dependent (25-10 points) and dependent (<10 points). The presence of functional decline was seen in those patients who had complete or partial dependence on IADL.
Assessment of biochemical determinations | Six months
  Venous blood samples were drawn from an antecubital vein early in the morning in a fasting state and assessed by a biochemical laboratory. The measured parameters included: Fasting plasma glucose (FPG), lipid profile (serum triglycerides _ TG, serum total cholesterol _ TC, serum low density lipoprotein cholesterol _ LDL-C, serum high density lipoprotein cholesterol _ HDL-C). Serum biochemistries were performed by automated enzimatic method, under routine laboratory procedures. The LDL-C was calculated using the Friedewald formula [22]. The normal values for parameters FPG, TG, TC, LDL-C, HDL-C used in this research were defined by the revised National Cholesterol Education Program (NCEP) Adult Treatment Panel III (ATP III).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil

REFERENCES:
- [Result] Kathiresan S, Otvos JD, Sullivan LM, Keyes MJ, Schaefer EJ, Wilson PW, D'Agostino RB, Vasan RS, Robins SJ. Increased small low-density lipoprotein particle number: a prominent feature of the metabolic syndrome in the Framingham Heart Study. Circulation. 2006 Jan 3;113(1):20-9. doi: 10.1161/CIRCULATIONAHA.105.567107. Epub 2005 Dec 27. PMID 16380547
- [Result] Hollenberg M, Yang J, Haight TJ, Tager IB. Longitudinal changes in aerobic capacity: implications for concepts of aging. J Gerontol A Biol Sci Med Sci. 2006 Aug;61(8):851-8. doi: 10.1093/gerona/61.8.851. PMID 16912104